CLINICAL TRIAL: NCT00106834
Title: A Phase 3, Multi-Center, Randomized, Double-Blind, Placebo-Controlled Trial Evaluating the Efficacy and Safety of Infliximab Induction and Maintenance Therapy in Patients With Moderate to Severe Plaque Psoriasis
Brief Title: A Study of the Safety and Efficacy of Infliximab in Patients With Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR003130
Record Dates: First submitted 2005-03-31; First posted 2005-04-01 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-03

CONDITIONS: Psoriasis
Keywords: Psoriasis; Infliximab; Remicade
MeSH Terms: conditions — Psoriasis | interventions — Infliximab

INTERVENTIONS:
Drug: Infliximab

SUMMARY:
The purpose of this study is to determine if infliximab (anti-TNF) is effective in the treatment of plaque psoriasis.

DETAILED DESCRIPTION:
This is an experimental medical research study. The purpose of this study is to determine if infliximab is effective in the treatment of plaque psoriasis. A total of about 375 patients primarily in Europe will participate in this study. The time of participation in this study is about 17 months. Infliximab is the active drug in Remicade. Infliximab is currently approved for the treatment of Crohn's disease (an irritable bowel disease), and rheumatoid arthritis. The usefulness and safety of infliximab in those diseases has been proven in previous research studies, which included more than 1300 patients in North America and Europe. In a previous small study of infliximab in 33 patients with psoriasis, about 80% of patients treated with infliximab showed improvement in their psoriasis symptoms after the first 3 infusions, while 20% of patients who received placebo showed improvement.

Patients will be assigned to one of two treatment groups (Group 1 and Group 2). Group 1 will receive 5mg/kg infliximab infusions at wks 0, 2, 4, 6, 14, 22, 30, 38 and 46 with placebo infusions at wks 24 and 26. Group 2 will receive placebo infusions at wks 0, 2, 6, 10, 14, 22, with placebo infusions at wks 24, 26, 30, 38 and 46. All study medication is given though an intravenous (into the vein) line.

Safety evaluations will be performed at specified intervals throughout the study and will consist of laboratory tests, vital signs (such as blood pressure), physical examinations and the occurrence and severity of adverse events as well as other study specific procedures. There are 2 different treatment groups: Group 1 will receive 5mg/kg infliximab infusions at wks 0, 2, 4, 6, 14, 22, 30, 38 and 46 with placebo infusions at wks 24 and 26. Group 2 will receive placebo infusions at wks 0, 2, 6, 10, 14, 22, with placebo infusions at wks 24, 26, 30, 38 and 46. All study medication is given though an intravenous (into the vein) line.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had a diagnosis of plaque-type psoriasis for at least 6 months
* Patients who have plaque-type psoriasis covering at least 10% of the body

Exclusion Criteria:

* Patients must not have nonplaque forms of psoriasis
* Patients must not have current drug-induced psoriasis
* Patients must not be pregnant, nursing, or planning pregnancy (both men and women) within 18 months of enrollment
* Patients must not have had any previous treatment with infliximab or any therapeutic agent targeted at reducing TNF

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving a = 75% improvement in Psoriasis Area and Severity Index (PASI) score from baseline at week 10

SECONDARY OUTCOMES:
The patients with = 75% improvement in PASI score from baseline to week 24 ,Change in Dermatology Life Quality Index from baseline to week 10 and week 24 , patients achieving a Physician Global Assessment score of cleared (0) or minimal(1) at week 10

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.

REFERENCES:
- [Background] Rich P, Griffiths CE, Reich K, Nestle FO, Scher RK, Li S, Xu S, Hsu MC, Guzzo C. Baseline nail disease in patients with moderate to severe psoriasis and response to treatment with infliximab during 1 year. J Am Acad Dermatol. 2008 Feb;58(2):224-31. doi: 10.1016/j.jaad.2007.07.042. Epub 2007 Dec 20. PMID 18083272
- [Result] Reich K, Nestle FO, Wu Y, Bala M, Eisenberg D, Guzzo C, Li S, Dooley LT, Griffiths CE. Infliximab treatment improves productivity among patients with moderate-to-severe psoriasis. Eur J Dermatol. 2007 Sep-Oct;17(5):381-6. doi: 10.1684/ejd.2007.0234. Epub 2007 Aug 2. PMID 17673380
- [Result] Reich K, Nestle FO, Papp K, Ortonne JP, Wu Y, Bala M, Evans R, Guzzo C, Li S, Dooley LT, Griffiths CE. Improvement in quality of life with infliximab induction and maintenance therapy in patients with moderate-to-severe psoriasis: a randomized controlled trial. Br J Dermatol. 2006 Jun;154(6):1161-8. doi: 10.1111/j.1365-2133.2006.07237.x. PMID 16704649
- [Result] Reich K, Nestle FO, Papp K, Ortonne JP, Evans R, Guzzo C, Li S, Dooley LT, Griffiths CE; EXPRESS study investigators. Infliximab induction and maintenance therapy for moderate-to-severe psoriasis: a phase III, multicentre, double-blind trial. Lancet. 2005 Oct 15-21;366(9494):1367-74. doi: 10.1016/S0140-6736(05)67566-6. PMID 16226614
- See also: A Phase 3, Multi-center, Randomized, Double-blind, Placebo-controlled Trial Evaluating the Efficacy and Safety of Infliximab Induction and Maintenance Therapy in Patients with Moderate to Severe Plaque Psoriasis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=143&filename=CR003130_CSR.pdf